CLINICAL TRIAL: NCT05706337
Title: Clinical Observation of Ciprofol for Anesthesia Induction in the Elderly Undergoing Elective Non-cardiac Surgery
Brief Title: Clinical Observation of Ciprofol for Anesthesia Induction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiumei Song (Other)
Responsible Party: Sponsor-Investigator, Xiumei Song, Associate chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YXLL-KY-2022(060)
Record Dates: First submitted 2022-11-29; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia; Pain; Hemodynamic Instability
Keywords: Anesthesia induction; Ciprofol; propofol; Injection pain
MeSH Terms: conditions — Pain | interventions — Propofol; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Active Comparator): According to grouping，patients were premeditated with injection of Propofol 1-2mg / kg IV . If BIS is ≤ 60, Tracheal intubation was facilitated with cisatracurium 0.2mg/kg a IV and sufentanil 0.3 μ g / kg IV. if BIS is >60, propofol 0.5mg/kg was titrated intravenously, with an interval of more than 1min until the BIS is ≤ 60，and intubation was performed after cisatracurium and sufentanil injected .General anesthesia was maintained with Propofol and remifentanil.
  Interventions: Drug: Propofol
- ciprofol group (Experimental): According to grouping，patients were premeditated with injection of ciprofol 0.2-0.5mg/kg IV. If BIS is ≤ 60, Tracheal intubation was facilitated with cisatracurium 0.2mg/kg a IV and sufentanil 0.3 μ g / kg IV. if BIS is >60, ciprofol 0.1mg/kg was titrated intravenously, with an interval of more than 1min until the BIS is ≤ 60，and intubation was performed after cisatracurium and sufentanil injected .General anesthesia was maintained with Propofol and remifentanil in both groups.
  Interventions: Drug: Ciprofol

INTERVENTIONS:
Drug: Propofol — Propofol 1-2mg / kg was for anesthesia induction. Propofol is a hypnotic agent that is used as an induction agent and as a maintenance anaesthetic delivered by continuous i.v. infusion or intermittent i.v. bolus.
  Arms: propofol group
Drug: Ciprofol — Ciprofol 0.2～0.5mg/kg was for anesthesia induction. Ciprofol is an intravenous sedative-hypnotic and a short-acting GABAA receptor agonist. It activates GABAergic neurons by enhancing chloride ion influx. It is used for anesthetic induction and maintenance agents include rapid induction of general anesthesia, rapid return of consciousness, minimal residual effects on the central nervous system and less injection pain.
  Arms: ciprofol group

SUMMARY:
To evaluate the effect of ciprofol anesthesia Induction on hemodynamics in elderly patients undergoing elective noncardiac surgery，a prospective, randomized, controlled trial.

DETAILED DESCRIPTION:
90 elderly patients undergoing noncardiac surgery were randomly divided into propofol group and ciprofol group, who were given propofol 1 ~ 2mg/kg or ciprofol 0.2-0.5mg/kg during anesthesia induction respectively. Systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR) and BIS values at various time points during anesthesia induction were collected. At the same time, rates of injection pain, muscle fasciculation, arrhythmia, cough and perioperative hepatic and renal functions were compared between the two groups. The primary outcomes were the fluctuations in hemodynamic parameters during induction. The secondary outcome were adverse reactions, BIS values and changes of hepatic and renal functions during induction.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status Ⅰ-Ⅲ
2. Age over 65 years;
3. Body mass index (BMI) 20 ~ 30 kg/m2 ;
4. Elective noncardiac surgery;

Exclusion Criteria:

1. The patient or his/her family refused to participate in the clinical trial;
2. Severe heart, lung, liver or kidney dysfunction;
3. Expected difficult airway, requiring awake tracheal intubation;
4. Those who are allergic to the drugs used in this study;
5. Unsuccessful tracheal intubation twice;
6. Patients with mental illness or impaired consciousness;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic changes：Systolic blood pressure (SBP) | From the beginning of drug administration to 30 minutes after intubation
  Systolic blood pressure (SBP) during anesthesia induction
Hemodynamic changes: Diastolic blood pressure(DBP) | From the beginning of drug administration to 30 minutes after intubation
  Diastolic blood pressure(DBP) during anesthesia induction
Hemodynamic changes: Heart rate （HR ） | From the beginning of drug administration to 30 minutes after intubation
  Heart rate （HR ）during anesthesia induction

SECONDARY OUTCOMES:
adverse reactions: injection pain | anesthesia induction
  injection pain from propofol or ciprofol intravenous injection
adverse reactions: muscle fasciculation | anesthesia induction
  muscle fasciculation induced by propofol or ciprofol intravenous induction
adverse reactions：arrhythmia | anesthesia induction
  arrhythmia induced by propofol or ciprofol intravenous induction
perioperative hepatic function: Aspartate Aminotransferase ( AST) | Before surgery , 1day after operation
  level of Aspartate Aminotransferase ( AST)
perioperative hepatic function: Alanine Aminotransferase ( ALT) | Before surgery , 1day after operation
  level of Alanine Aminotransferase ( ALT)
perioperative renal function: creatine | Before surgery , 1day after operation
  level of creatine
perioperative renal function:Blood Urea Nitrogen | Before surgery , 1day after operation
  level of Blood Urea Nitrogen（BUN)
Monitoring Depth of Anesthesia | anesthesia induction
  BIS values

CONTACTS AND LOCATIONS:
Overall Officials: Xiumei Song, Doctor, Study Chair — Qian fo shan hospitial of shan dong province, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to upload and share data with other researchers. Protecting patient privacy when sharing patient-level data from clinical trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: study protocol and Informed Consent Form will available before 2024/1/1 Statistical Analysis Plan and Clinical Study Report will available before 2024/6/1
Access Criteria: All registered researchers

REFERENCES:
- [Background] Teng Y, Ou M, Wang X, Zhang W, Liu X, Liang Y, Li K, Wang Y, Ouyang W, Weng H, Li J, Yao S, Meng J, Shangguan W, Zuo Y, Zhu T, Liu B, Liu J. Efficacy and safety of ciprofol for the sedation/anesthesia in patients undergoing colonoscopy: Phase IIa and IIb multi-center clinical trials. Eur J Pharm Sci. 2021 Sep 1;164:105904. doi: 10.1016/j.ejps.2021.105904. Epub 2021 Jun 8. PMID 34116176
- [Background] Wang X, Wang X, Liu J, Zuo YX, Zhu QM, Wei XC, Zou XH, Luo AL, Zhang FX, Li YL, Zheng H, Li H, Wang S, Wang DX, Guo QL, Liu CM, Wang YT, Zhu ZQ, Wang GY, Ai YQ, Xu MJ. Effects of ciprofol for the induction of general anesthesia in patients scheduled for elective surgery compared to propofol: a phase 3, multicenter, randomized, double-blind, comparative study. Eur Rev Med Pharmacol Sci. 2022 Mar;26(5):1607-1617. doi: 10.26355/eurrev_202203_28228. PMID 35302207
- [Background] Qin K, Qin WY, Ming SP, Ma XF, Du XK. Effect of ciprofol on induction and maintenance of general anesthesia in patients undergoing kidney transplantation. Eur Rev Med Pharmacol Sci. 2022 Jul;26(14):5063-5071. doi: 10.26355/eurrev_202207_29292. PMID 35916802
- See also: Liu J, Wang D , Zuo Y, MI W, Yao S, Yu W. Guidelines on clinical application of ciprofol. Chin J Anesthesiol, 2021,41 (2): 129-132 — http://rs.yiigle.com/CN131073202102/1326216.htm